CLINICAL TRIAL: NCT07138638
Title: High-Frequency QRS for Predicting Microvascular Dysfunction and Adverse Events After PCI in Acute Myocardial Infarction: A Prospective, Multicenter Cohort Study
Brief Title: High-Frequency QRS for Predicting Microvascular Dysfunction and Adverse Events After PCI in Acute Myocardial Infarction
Status: Not yet recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: XYFY2025-KL303-01
Record Dates: First submitted 2025-08-13; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: AMI
Keywords: Acute Myocardial Infarction; High-Frequency QRS; prediction model; Microvascular Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: High-Frequency QRS — All enrolled patients underwent HF-QRS assessment, with subsequent recording of MACE to evaluate the predictive value of HF-QRS parameters for clinical outcomes

SUMMARY:
This observational study aimed to investigate the prognostic value of high-frequency QRS (HF-QRS) in patients with acute myocardial infarction (AMI) after percutaneous coronary intervention (PCI), as well as its potential role in diagnosing microvascular dysfunction. The main question it aims to answer is:

1. Whether HF-QRS could serve as an effective tool for early identification of high-risk AMI patients and prognosis prediction;
2. Whether HF-QRS provides auxiliary diagnostic value for post-AMI microvascular dysfunction.

Participants underwent HF-QRS assessment and were prospectively followed for 1 year to record the incidence of major adverse cardiovascular events (MACE).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years (inclusive)

Diagnosed with acute myocardial infarction (AMI, including STEMI and NSTEMI) and underwent successful emergency PCI

Voluntarily participated and provided written informed consent

Exclusion Criteria:

* History of prior myocardial infarction or chronic heart failure

QRS duration >120 ms (including paced rhythm, WPW syndrome, bundle branch block, or left ventricular hypertrophy with repolarization abnormalities)

Structural heart disease (congenital heart disease, cardiomyopathy, aortic dissection, etc.)

Persistent atrial fibrillation or malignant arrhythmias

History of cerebral hemorrhage or ischemic stroke within 1 month

Prolonged cardiopulmonary resuscitation or requiring advanced life support (IABP/ECMO, etc.)

Scheduled for imminent surgery with anticipated inability to complete HF-QRS assessment

Other life-threatening conditions including: Severe hepatic or renal dysfunction;Uncontrolled systemic diseases;Hematologic disorders;Active infections;Malignancy with life expectancy <1 year Other investigator-determined exclusionary conditions:Pregnancy;Concurrent participation in other clinical trials

Refusal to participate in the clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute myocardial infarction following percutaneous coronary intervention
Sampling Method: Probability Sample
Enrollment: 1112 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the predictive value of high-frequency QRS (HF-QRS) parameters for major adverse cardiovascular events (MACE) within 1 year after PCI in AMI patients and to construct a prognostic risk prediction model. | 12 months

SECONDARY OUTCOMES:
To evaluate the adjunctive diagnostic value of high-frequency QRS parameters for microvascular dysfunction in ACS patients following percutaneous coronary intervention | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, Ph.D, Study Chair — Department of Cardiology, Peking University First Hospital, Beijing, China; Yuan Lu, Ph.D, Study Director — The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu 221002
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No